CLINICAL TRIAL: NCT00006015
Title: Phase II Study Evaluating the Combination of 5-Fluorouracil, Leucovorin, Oxaliplatin, and Herceptin in the Treatment of Patients With Metastatic Colorectal Cancer Who Have Progressed After 5-FU and/or Irinotecan-Containing Therapy
Brief Title: Combination Chemotherapy Plus Trastuzumab in Treating Patients With Advanced, Recurrent, or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of sufficient accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Monica M Bertagnolli, Cancer and Leukemia Group B
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068024; U10CA031946 (NIH); CALGB-89902
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Trastuzumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Chemotx (Experimental): Combination chemotherapy for metastatic colorectal cancer in patients who have disease progression after 5-FU and/or irinotecan-containing therapy
  Interventions: Biological: trastuzumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: trastuzumab — 4 mg/kg IV infusion Day 1, then weekly 2 mg/kg IV infusion (on Days 8, 15, & 22)
  Other Names: Herceptin
Drug: fluorouracil — 500 mg/sq m IV push weekly for 3 weeks, followed by a 1 wk break
  Other Names: 5-FU
Drug: leucovorin calcium — 500 mg/sq m IV infusion over 2 hours weekly for 3 weeks, then a 1 wk break
Drug: oxaliplatin — 85 mg/sq m IV infusion over 2 hours Days 1 & 15 of each cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying combination chemotherapy plus trastuzumab to see how well it works in treating patients with advanced, recurrent, or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients who overexpress HER-2/neu with metastatic colorectal adenocarcinoma who have progressed on at least 1 prior, but no more than 2 prior, chemotherapy regimens for metastatic colorectal cancer treated with fluorouracil, leucovorin calcium, oxaliplatin, and trastuzumab (Herceptin).
* Determine the time to progression of these patients treated with this regimen.
* Determine the overall toxicity of this regimen in these patients.

OUTLINE: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22, followed by oxaliplatin IV over 2 hours on days 1 and 15, and then followed by leucovorin calcium IV over 2 hours on days 1, 8, and 15. Fluorouracil IV is administered at the midpoint of the leucovorin calcium infusion on days 1, 8, and 15. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 20-45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced, recurrent, or metastatic colorectal adenocarcinoma
* Resected CNS metastases stable greater than 1 month after completion of radiotherapy for CNS metastases eligible

  * No existing CNS metastases allowed
* Measurable disease

  * At least 1 dimension as at least 20 mm with conventional techniques OR
  * At least 10 mm with spiral CT scan
  * No truly nonmeasurable lesions:

    * Bone lesions
    * Leptomeningeal disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Must have progressed on at least 1 prior, but no more than 2 prior, fluorouracil and/or irinotecan containing treatment regimens for metastatic colorectal cancer
* Must have documented HER-2/neu overexpression by immunohistochemistry staining

  * Staining score at least 2+

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of cardiac ischemia or congestive heart failure
* LVEF at least 50% by ECG or MUGA

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent second malignancy except nonmelanoma skin cancers or carcinoma in situ of the cervix unless completed therapy and considered to be at less than 30% risk of relapse

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior platinum containing chemotherapy
* At least 3 weeks since prior chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-05; Primary Completion 2002-12 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 2 tx cycles
Time to progression | Every 2 tx cycles
Overall toxicity | Each cycle during tx

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Clark, MD, Study Chair — Massachusetts General Hospital
Locations (47):
- United States (47):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Clark JW, Niedzwiecki D, Hollis D, et al.: Phase II trial of 5-fluororuacil (5-FU), leucovorin (LV), oxaliplatin (Ox), and trastuzamab (T) for patients with metastatic colorectal cancer (CRC) refractory to initial therapy. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3584, 2003.